CLINICAL TRIAL: NCT04440371
Title: Comparison of the Efficacy of Tacrolimus 0.1% Ointment vs Calcipotriol/Betamethasone in Combination With NBUVB in Treatment of Vitiligo
Brief Title: Phototherapy Combination With Topicals in Vitiligo
Acronym: NBUVB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/104/2017
Record Dates: First submitted 2020-05-28; First posted 2020-06-19 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Vitiligo, Generalized
MeSH Terms: conditions — Vitiligo | interventions — Tacrolimus; calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus (Active Comparator): Phototherapy NBUVB will be given 3 times per week and Tacrolimus 0.1% ointment will be applied twice a day
  Interventions: Combination Product: Tacrolimus 0.1% ointment twice daily plus NBUVB 3 times weekly; Combination Product: Calcipotriol/Betamethasone ointment plus NBUVB
- calcipotriol / betamethasone (Active Comparator): Phototherapy NBUVB will be given 3 times per week and calcipotriol & betamethasone containing cream will be applied once a day
  Interventions: Combination Product: Tacrolimus 0.1% ointment twice daily plus NBUVB 3 times weekly; Combination Product: Calcipotriol/Betamethasone ointment plus NBUVB

INTERVENTIONS:
Combination Product: Tacrolimus 0.1% ointment twice daily plus NBUVB 3 times weekly — Tacrolimus ointment plus phototherapy NBUVB (Tacrolimus arm)
Combination Product: Calcipotriol/Betamethasone ointment plus NBUVB — Calcipotriol/Betamethasone ointment once daily plus NBUVB 3 times weekly

SUMMARY:
Patients will be included in a randomized controlled clinical trial, will enroll only adult vitiligo patients with surface area of at least 10% who are being followed in the outpatient dermatology clinics of King Abdullah University Hospital (KAUH) and are planned to start on phototherapy Narrow Band Ultraviolet light B (NBUVB), regardless if they have previous treatment for their disease, one month wash off period will be given for patients who are already on phototherapy or other treatments for vitiligo.

DETAILED DESCRIPTION:
Patients to be included in this randomized controlled study are adults with generalized vitiligo of surface area of at least 10% who are being followed in the outpatient dermatology clinics of King Abdullah University Hospital (KAUH) and are planned to start on phototherapy Narrow Band Ultraviolet light B (NB-UVB), regardless if they have previous treatment for their disease, one month wash off period will be given for patients who are already on phototherapy or other treatments for vitiligo. In our going study, adult patients will be enrolled into 2 groups ( around 20 patients per each) in which NBUVB will be given 2-3 sessions per week in combination with one of the following randomly; one group will start on Tacrolimus 0.1% ointment twice daily, a second group will start on calcipotriol & betamethasone containing cream once daily, photos will be taken and the exact sites involved will be detected, efficacy of treatment will be assessed according to repigmentation percentages of vitiligo areas from baseline at 3 and 6 months. The improvement at 6 months compared to baseline will be classified into 5 groups according to the percentage of repigmentation as follow; excellent (76%-100%); moderate (51%-75%); mild (26%-50%); minimal (1%-25%); or no response.

ELIGIBILITY:
Inclusion criteria:

* Adult patients ( ≥ 18 years).
* Diagnosed with vitiligo clinically and by using wood's light
* Generalized type vitiligo and BSA ≥ 10%
* Planned by his physician to start on phototherapy
* Wash off period for patients on treatment of one month duration.

Exclusion criteria:

* Children less than 18 year old
* Localized type vitiligo or BSA less than 10%
* Unable to do phototherapy
* Pregnant women with vitiligo
* Previously failed to response to phototherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-21 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
efficacy of treatment | Baseline: measurement of vitiligo BSA with photographs of vitiligo areas. lab investigations done at this stage
  The area of vitiligo will be measured using body surface area (BSA) at baseline. the difference in BSA will represent the improvement from baseline. Patient palm will be used for estimation of BSA at each visit (Each one plam is equivalent to 1% of BSA). Photographs will be taken .
Efficacy of treatment | 3 months post treatment
  The area of vitiligo will be measured using body surface area (BSA) at 3 months. the difference in BSA will represent the improvement from baseline. Patient palm will be used for estimation of BSA at each visit (Each one plam is equivalent to 1% of BSA). Photographs will be taken.
Efficacy of treatment | 6 months post treatment
  The area of vitiligo will be measured using body surface area (BSA). the difference in BSA will represent the improvement from baseline. Patient palm will be used for estimation of BSA at each visit (Each one plam is equivalent to 1% of BSA). Photographs will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Diala Alshiyab, MD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Diala Alshiyab, Irbid, Jordan

REFERENCES:
- [Derived] Alshiyab D, Al-Qarqaz F, Ba-Shammakh S, Al-Fakih A, Altawalbeh A, Alsheyab S, Sarakbi D, Muhaidat J. Comparison of the efficacy of tacrolimus 0.1% ointment vs calcipotriol/betamethasone in combination with NBUVB in treatment of vitiligo. J Dermatolog Treat. 2023 Dec;34(1):2252119. doi: 10.1080/09546634.2023.2252119. PMID 37644869